CLINICAL TRIAL: NCT02911363
Title: Randomized Trial Comparing Captivator Tissue Cassettes vs. no Cassettes for Endoscopic Mucosal Resection in Esophageal Carcinoma
Brief Title: Comparison of Captivator Tissue Cassettes vs. no Cassettes for Endoscopic Mucosal Resection in Esophageal Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 724207
Record Dates: First submitted 2016-04-12; First posted 2016-09-22 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capitvator Cassette (Active Comparator): The EMR specimen will be processed using the Captivator Cassette.
  Interventions: Device: Captivator cassette
- Standard of Care Processing (Active Comparator): The EMR specimen will be prepared per Standard of Care.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Captivator cassette — The Captivator tissue cassette has an effect on the preservation of tissue histology.
  Arms: Capitvator Cassette
Other: Standard of Care — The specimen will be processed following the College of American Pathology Standards.
  Arms: Standard of Care Processing

SUMMARY:
The main purpose of this study will be to two-fold; firstly to determine whether the use of a Captivator tissue cassette has an effect on the preservation of tissue histology (minimizing artifactual curling) , and secondly to determine whether the use of a intraprocedural cassette is practical. The investigators believe that this will greatly aid in elucidating the best technique for optimizing performance of EMR for esophageal lesions.

DETAILED DESCRIPTION:
As a result of the advances in endoscopic procedures, the detection of early stage esophageal carcinoma has increased. Endoscopic mucosal resection (EMR) is an innovative technique for removal of high grade intraepithelial neoplasia/dysplasia to prevent the progression of invasive carcinoma which occurs in about a third of patients. EMR involves the endoscopic therapeutic removal of the abnormal esophageal area(s) of tissue by snare or suction, aiming to include as much of the submucosal layer as possible, which is (are) then submitted for histopathological examination for pathological diagnosis and tumor staging. Compared with esophageal biopsy, this methodology reveals more advanced tumor stages in terms of grading and vertical infiltration in 10-20% of patients. Because of the importance of histopathologic diagnosis, the specimen should be pinned on a cork or styrofoam board to prevent curling and maintain the orientation, integrity of the size and shape, and fixed in an appropriate volume of 10% formalin. Unfortunately, specimens are often not pinned as EMR specimens can be difficult and time consuming to pin because of their thickness, hence the specimen integrity (size and shape) and orientation is compromised.

Therefore the main purpose of this study will be to two-fold; firstly to determine whether the use of a Captivator tissue cassette has an effect on the preservation of tissue histology (minimizing artifactual curling) , and secondly to determine whether the use of a intraprocedural cassette is practical. The investigators believe that this will greatly aid in elucidating the best technique for optimizing performance of EMR for esophageal lesions.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to Florida Hospital Endoscopy Unit for assessment of an esophageal lesion that require EMR
* Age ≥ 19 years

Exclusion Criteria:

* Age <19 years
* Unable to safely undergo EMR for any reason
* Coagulopathy (INR >1.6, Thrombocytopenia with platelet count <80,000/ml)
* Unable to provide consent for any reason
* Pregnancy (confirmed with Standard of Care urine pregnancy test for all women with child-bearing potential)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Histological quality of the EMR specimen obtained during the procedure will be analyzed and compared to cassette vs. no cassette for pathology review. | 1 year
  1. Captivator tissue cassette vs. no cassette
  1. Captivator tissue cassette with margin curling/artifact vs. Captivator tissue cassette without margin curling/artifact
  2. No cassette with margin curling/artifact vs. no cassette without margin curling/artifact
  3. Captivator tissue cassette with margin curling/artifact vs. No cassette with margin curling/artifact

SECONDARY OUTCOMES:
Ease of use of the Captivator tissue cassette will be comparable to Standard of Care. | 1 year
  Ease of use of the Captivator tissue cassette will be comparable in terms of handling the histologic specimen and will not add significant time to the intraprocedural or laboratory handling and processing.

CONTACTS AND LOCATIONS:
Overall Officials: Shantel Hebert-Magee, MD, Principal Investigator — Florida Hospital Orlando
Locations (1):
- Center for Interventional Endoscopy - Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2013. CA Cancer J Clin. 2013 Jan;63(1):11-30. doi: 10.3322/caac.21166. Epub 2013 Jan 17. PMID 23335087
- [Background] Devesa SS, Blot WJ, Fraumeni JF Jr. Changing patterns in the incidence of esophageal and gastric carcinoma in the United States. Cancer. 1998 Nov 15;83(10):2049-53. PMID 9827707
- [Background] Blot WJ, McLaughlin JK. The changing epidemiology of esophageal cancer. Semin Oncol. 1999 Oct;26(5 Suppl 15):2-8. PMID 10566604
- [Background] Lagergren J, Bergstrom R, Lindgren A, Nyren O. Symptomatic gastroesophageal reflux as a risk factor for esophageal adenocarcinoma. N Engl J Med. 1999 Mar 18;340(11):825-31. doi: 10.1056/NEJM199903183401101. PMID 10080844